CLINICAL TRIAL: NCT02011074
Title: Perioperative Changes of Heart Rate Variability Related to Anxiety and Depressiveness in Psychologically Normal Patients Undergoing General Anesthesia
Brief Title: Perioperative Changes of Heart Rate Variability Related to Anxiety and Depressiveness in Patients Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung Hee Kim, MD. PhD, Samsung Medical Center
Other Study IDs: 2012-08-043
Record Dates: First submitted 2013-11-28; First posted 2013-12-13 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Heart Rate Variability; STAI; SDS; General Anesthesia; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Preoperative anxiety can be detected via structured and standardised screening by the State - Trait Anxiety Inventory (STAI) and Self rating Depression Scale (SDS) questionnaire. The investigators evaluate the relation of perioperative anxiety and heart rate variability, also the impact of general anesthesia on the change of heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma patients

Exclusion Criteria:

* uncontrolled hypertension uncontrolled diabetes mellitus known autonomic nerve dysfunction

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatocellular carinoma patients undegoing Hepatectomy with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | change from baseline in HRV at 10 minutes after induction of general anesthesia

SECONDARY OUTCOMES:
STAI score | change from baseline in HRV at 10 minutes after induction of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Kim Myunghee, Gangnamgu, Seoul, South Korea